CLINICAL TRIAL: NCT00638430
Title: The Effect of Myopic Optical Defocus on the Humphrey Matrix 30-2 Test
Status: Completed | Type: Observational
Sponsor: Samsung Medical Center (Other)
Responsible Party: Changwon Kee, Department of Ophthalmology, Samsung Medical Center,
Other Study IDs: Humphrey30-2
Record Dates: First submitted 2008-03-12; First posted 2008-03-19 (Estimated); Last update posted 2008-03-19 (Estimated); Status verified 2008-03

CONDITIONS: Myopia
Keywords: myopia; Humphery Matrix 30-2 test
MeSH Terms: conditions — Myopia

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (2):
- 1: low myopic group
- 2: moderate myopic group

SUMMARY:
The purpose of this study is to examine the effect of the myopic optical defocus on the Humphrey Matrix 30-2 test.

DETAILED DESCRIPTION:
The Humphery Matrix (Zeiss, Dublin, California, USA; in cooperation with Welch Allyn, Skaneateles, New York, USA), which is a recently developed version of FDT perimetry, showed more improved technology to detect early glaucomatous damage. The user's guide for the Humphrey Matrix (Humphrey® matrix visual field instrument user's guide. Zeiss, Dublin, California, USA; in cooperation with Welch Allyn, Skaneateles, New York, USA; 2003) suggests that myopic refractive errors more than -3.0 D need to be corrected before the 30-2 test. However, the proper correction of the optical defocus is not always easy because of a lack of trial frame.

The purpose of the present study is twofold. At first, the influence of the low-grade myopia on the Humphery Matrix 30-2 test will be evaluated and compared to the effect of moderate-grade myopia. Secondly, the influence of myopic optical defocus and the glaucomatous visual field damage on the pattern deviation plot change according to the severity of glaucomatous visual field damage will be estimated.

ELIGIBILITY:
Inclusion Criteria:

* intra-ocular pressure 23 or higher
* suspicious glaucomatous optic disc change
* suspicious defect of retinal nerve fiber layer
* or eyes with various degrees of glaucoma

Exclusion Criteria:

* a high myopic eye (SE more than -6.0 D)
* moderate to severe cataract
* evidence of diabetic or hypertensive retinopathy
* macular disease
* intra-ocular inflammation
* history of intraocular surgery and any other ocular lesion that could have an influence on the perimetry result

Ages: 27 Years to 61 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Study Population: tertiary care clinic
Sampling Method: Non-Probability Sample
Enrollment: 40 (Actual)
Dates: Start 2007-03; Primary Completion 2007-10 (Actual); Study Completion 2008-03 (Actual)

PRIMARY OUTCOMES:
mean defect | 15 minutes

CONTACTS AND LOCATIONS:
Overall Officials: Changwon Kee, M.D., Study Chair — Department of Ophthalmology, Samsung Medical Center,
Locations (1):
- Samsung Medical Center, Seoul, South Korea

REFERENCES:
- [Result] Anderson AJ, Johnson CA. Frequency-doubling technology perimetry and optical defocus. Invest Ophthalmol Vis Sci. 2003 Sep;44(9):4147-52. doi: 10.1167/iovs.02-1076. PMID 12939339